CLINICAL TRIAL: NCT02176681
Title: A Prospective, Multicenter, Randomized, Open-label Study of 12 Week Duration to Evaluate the Effect of VILDagliptin Added to Insulin on Glycaemic Control in haemoDIALyzed Patients With Type 2 Diabetes: Probe Analysis of CGM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5706
Record Dates: First submitted 2014-06-05; First posted 2014-06-27 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Haemodialyzed, Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin alone (Active Comparator): Use the usual frequency and dose
  Interventions: Drug: Insulin
- Insulin and Vildagliptin (Experimental): vildagliptin 50 mg/day during 3 months

INTERVENTIONS:
Drug: Vildagliptin (Galvus) — Use Vildagliptin (50 mg/day) added to insulin during 3 months
Drug: Insulin — Insulin
  Arms: Insulin alone

SUMMARY:
Diabetes is a major concern for dialysis units, as it is now the most common cause of end-stage renal disease in France. In 2010 at initiation of dialysis treatment, more than one patient out of two had at least one cardiovascular disease and 40 % diabetes (94 % Type 2 diabetes) and especially in East part of France.

Diabetic patients on dialysis have a high burden of morbidity and mortality, particularly from cardiovascular disease. Tight glycaemic and blood pressure control in diabetic patients has an important impact in reducing risk of progression nephropathy. Data are scarce on how diabetes should best be treated in dialysis patients. The evidence for improving glycaemic control in patients on dialysis having an impact on mortality or morbidity is sparse. Indeed, many factors make improving glycaemic control in patients on dialysis very challenging, including therapeutic difficulties with hypoglycaemic agents, monitoring difficulties, dialysis strategies that exacerbate hyperglycaemia or hypoglycaemia.

Standard oral drugs therapy for hyperglycaemia (eg, metformin, sulfonylureas, ) are contraindicated in patients on dialysis. Thus insulin has been the mainstay of treatment. Newer therapies for hyperglycaemia, such as gliptins and glucagon-like peptide-1 analogues have become available, but until recently, renal failure has precluded their use. Newer gliptins, however, are now licensed for use in 'severe renal failure', although they have yet to be trialed in dialysis patients.

The investigators study, using continuous glucose monitoring as a new tool for monitoring of therapy should provide information on vildagliptin in add on therapy to insulin in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by haemodialysis for more than 3 months with 1g/L glucose in dialysate fluid
* Patients treated by stable doses of insulin (any regimen) for Type 2 diabetes without any oral antidiabetic agent
* Age > 18 years
* TGO, TPO and lipase < 3x ULN
* effective means of contraception

Non-inclusion Criteria:

* Blood transfusion in the 2 previous months
* Life expectancy less than 1 year
* Chronic inflammatory disease
* Steroid treatment > 5mg/day
* Cancer (evolutive or requiring chemotherapy or radiotherapy) with the exception of breast intraductal carcinoma operated
* Patient waiting for programmed surgery
* History of cardiovascular disease (stroke, coronary heart disease, hospitalization for heart failure) in the 4 previous months
* Patients suffering from stage 3 and 4 cardiac insufficiency
* Non-compliant patients
* History of pancreatitis
* History of angioedema
* Hypersensitivity to the active substance or to any of the excipients of Galvus®
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Mean glucose value of CGM [M] to be averaged from day 2 and day 3 of CGM | up to day 3

SECONDARY OUTCOMES:
CGM parameters at baseline and month 3 | Other CGM parameters at baseline and month 3
  glucose area under the curve (AUC) for glucose value higher than 7.7 mmol/l
  * number of glucose values under 3.3 mmol/l
  * hypoglycaemic events at baseline, month 3
  * number of minor hypoglycaemic events per month
  * number of major hypoglycaemic events at month 3
  * number of nocturnal hypoglycaemic events per month
  * variability glycemic index: MAGE, CV
Number of hypoglycaemic events | Hypoglycaemic events at baseline, month 3
  hypoglycaemic events at baseline, month 3
  * number of minor hypoglycaemic events per month
  * number of major hypoglycaemic events at month 3
  * number of nocturnal hypoglycaemic events per month
Mean HbA1C and Glycated albumin | HbA1C and Glycated albuminat baseline and month 3

CONTACTS AND LOCATIONS:
Overall Officials: François CHANTREL, MD, Principal Investigator — AURAL - Mulhouse; Alexandre KLEIN, MD, Principal Investigator — Hospices Civils de Colmar; Olivier IMHOFF, MD, Principal Investigator — AURAL Clinique Saint-Anne de Strasbourg; Alexandre KLEIN, MD, Principal Investigator — AURAL - Colmar; Dominique FLEURY, MD, Principal Investigator — CH de Valenciennes; Bruno VERGES, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Philippe ZAOUI, MD-PhD, Principal Investigator — University Hospital, Grenoble; Philippe ZAOUI, MD-PH, Principal Investigator — AGDUC - Grenoble; Gabriel CHOUKROUN, MD PhD, Principal Investigator — Centre Hospitalier Universitaire, Amiens; Joëlle CRIDLIG, MD, Principal Investigator — Central Hospital, Nancy, France; Sophie BOROT, MD, Principal Investigator — CHU de Besançon; François CHANTREL, MD, Principal Investigator — CH de Mulhouse; Olivier IMHOFF, MD, Principal Investigator — Clinique Sainte Anne de Strasbourg; Kristian KUNTZ, MD, Principal Investigator — AURAL de Strasbourg
Locations (13):
- France (13):
  - CH d'Amiens, Amiens
  - CH de Besançon, Besançon
  - AURAL Colmar, Colmar
  - Hospices civils de Colmar, Colmar
  - CH de Dijon, Dijon
  - AURAL Mulhouse, Mulhouse
  - CH de Mulhouse, Mulhouse
  - CH de Nancy, Nancy
  - AURAL Clinique Sainte Anne, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - AURAL Strasbourg, Strasbourg
  - CH de Valenciennes, Valenciennes

REFERENCES:
- [Result] Munch M, Meyer L, Hannedouche T, Kunz K, Alenabi F, Winiszewski P, Baltzinger P, Smagala A, Klein A, Dorey F, Fleury D, Verier-Mine O, Guerci B, Cridlig J, Borot S, Ducloux D, Meyer N, Hadjadj S, Chantrel F, Kessler L. Effect of adding vildagliptin to insulin in haemodialysed patients with type 2 diabetes: The VILDDIAL study, a randomized, multicentre, prospective study. Diabetes Obes Metab. 2020 Jun;22(6):978-987. doi: 10.1111/dom.13988. Epub 2020 Feb 25. PMID 32048396